CLINICAL TRIAL: NCT05548153
Title: An Observational Study on the Relationship Between Tear Metabolomics and POD
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: tear and delirium
Record Dates: First submitted 2022-09-06; First posted 2022-09-21 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tear was collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the correlation between tear metabolomics and POD. The purpose of this study was to compare the results of tear metabolomics between POD and non-POD elderly patients undergoing abdominal surgery, to clarify the correlation between tear metabolomics and POD, and to find tear markers related to POD.

ELIGIBILITY:
Inclusion Criteria:

* age 65-90 years old;
* ASA I-III;
* patients who plan to undergo elective abdominal surgery under general anesthesia;
* Volunteer to participate in this study and sign informed consent.

Exclusion Criteria:

* patients with known mental illness or lack of communication or cognitive impairment before operation;
* severe vision, hearing, language impairment or other reasons unable to communicate with visitors;
* severe dysfunction of important organs such as heart, brain, lung, liver, kidney, etc.;
* long-term use of sedatives, antidepressants or alcoholism;
* patients with severe postoperative complications and admitted to intensive care unit;
* patients who refused or failed to complete the cognitive function test.
* patients who could not cooperate with the study for any other reason

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: In the elderly patients who underwent abdominal surgery under general anesthesia, there were no serious systemic diseases and severe cognitive impairment before operation.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium during the 3 adys-follow-up after anesthetic resuscitation | From ending of the surgery to 3 days after anesthetic resuscitation
  Postoperative delirium was tested with 3D-Confusion Assessment Method or Confusion Assessment Method-intensive care unit (0-4, higher scores means worse). The patient is determined to be postoperative delirium (ie, Confusion Assessment Method positive) if he/she fall ill quickly with confusion disorder, and with mental disorder or consciousness disorder.

SECONDARY OUTCOMES:
Postoperative delirium in the postanesthesia care unit | From ending of the surgery to the time when discharge from postanesthesia care unit, an average of 30 minutes.
  Postoperative delirium was tested with Confusion Assessment Method-intensive care unit. Postoperative delirium was tested with Confusion Assessment Method-intensive care unit (0-4, higher scores means worse outcome). The patient is determined to be postoperative delirium (ie, Confusion Assessment Method positive) if he/she fall ill quickly with confusion disorder, and with mental disorder or consciousness disorder.
Postoperative delirium on the first day after operation | 9：00-10：00 and 15：00-16：00 on The first day after operation
  Postoperative delirium was tested with 3D-Confusion Assessment Method (0-4, higher scores means worse outcome). The patient is determined to be postoperative delirium (ie, Confusion Assessment Method positive) if he/she fall ill quickly with confusion disorder, and with mental disorder or consciousness disorder.
Postoperative delirium on the second day after operation | 9：00-10：00 and 15：00-16：00 on The second day after operation
  Postoperative delirium was tested with 3D-Confusion Assessment Method (0-4, higher scores means worse outcome). The patient is determined to be postoperative delirium (ie, Confusion Assessment Method positive) if he/she fall ill quickly with confusion disorder, and with mental disorder or consciousness disorder.
Postoperative delirium on the third day after operation | 9：00-10：00 and 15：00-16：00 on The third day after operation
  Postoperative delirium was tested with 3D-Confusion Assessment Method (0-4, higher scores means worse outcome). The patient is determined to be postoperative delirium (ie, Confusion Assessment Method positive) if he/she fall ill quickly with confusion disorder, and with mental disorder or consciousness disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Huang He, MD, Study Director — Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email
Supporting Information: Study Protocol, SAP, ICF, CSR